CLINICAL TRIAL: NCT06857864
Title: Exploratory Study on the Effectiveness of Myopia Control Lenses in Slowing Myopia Progression in Young Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WS10441
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Myopia
Keywords: Myopia; Refractive errors; Eye Diseases
MeSH Terms: conditions — Myopia; Refractive Errors; Eye Diseases

STUDY DESIGN:
Intervention Model Description: This is a mono-center, single-arm, unmasked study consisting of 6 visits over 1 year. This study aims to evaluate the change in axial elongation and spherical equivalent refraction in younger children who are fitted with the test lenses over a 1-year period.
  After obtaining informed consent and assent, a comprehensive eye examination will be conducted during the screening visit on all participants. Eligible participants, total of 25, between ages 6 to 8 years old will be enrolled into the study. On a separate visit, the enrolled subjects will return for a baseline visit to collect the study spectacles. During the baseline visit, instructions on study spectacles usage, assessment with study spectacles and ocular biometry will be conducted. Follow-up visits will be conducted at 3, 6 and 12 months' time, where 12 months is the end of study.
  All eye examinations and assessments are non-contact and non-invasive to the eyes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test myopia control lenses (BSL) (Experimental): Test spectacle lens will be given to the subjects over 1 year.
  Interventions: Device: Test myopia control lenses (BSL)

INTERVENTIONS:
Device: Test myopia control lenses (BSL) — Test spectacle lenses will be provided to the subjects throughout the 1 year clinical trial.

SUMMARY:
This study will be a mono-center, single-arm, unmasked study evaluating the effectiveness of test lens in slowing myopia progression in children aged 6 to 8 years. The study aims to evaluate the change in axial elongation and spherical equivalent refraction in younger children who are fitted with the test lens over a 1-year period. A total of 25 children will be recruited.

DETAILED DESCRIPTION:
As myopia has become a global epidemic and public health concern, it is crucial to gain deeper insight to the possible treatments in slowing myopia progression. In a previous clinical trial, spectacle lenses with higher lenlets asphericity demonstrated effectiveness in reducing myopia progression and axial length elongation in children.

This clinical trial will assess the effectiveness of a test lens in slowing myopia progression in younger children over 1 year. Without compromising vision, the test lens is designed to modify the area and the amount of myopia defocus on the retina. The study population includes 25 children subjects in Singapore, aged 6 to 8 years during the commencement of the treatment. The axial length and spherical equivalent refraction will be the primary and secondary measures for myopia progression.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer subject and guardian, fluent English spoken, willing to follow protocol and able to read, comprehend and sign the informed consent & assent form.
* Equal to or greater than 6 years and less than 9 years at time of informed consent and assent.
* Spherical equivalent refractive error (SER) by manifest refraction between -0.75 and -4.75 D in each eye.
* Astigmatism, if present, of not more than 1.50 D.
* Difference in SER between the two eyes (Anisometropia) by manifest refraction not more than 1.00 D.
* Best corrected visual acuity in each eye equal to or better than +0.10 logMAR (≥ 20/25 as Snellen)
* Be in good general health based on his/her and parent's/guardian's knowledge. Absence of ocular disease with full ophthalmic examination. Without any ocular or systemic condition known to affect refractive status.
* Absence of strabismus by cover test at near or distance wearing correction.
* Absence of amblyopia
* Without ocular or systemic medications which, in the investigator's opinion, may significantly affect pupil size, accommodation or refractive state.

Exclusion Criteria:

* Vulnerability of subject
* History of myopia control intervention
* Participation in any clinical study within 30 days of the Baseline visit.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Axial length | 12 months
  Evaluate the change in axial length (mm)

SECONDARY OUTCOMES:
Axial length | 6 months
  Evaluate change in axial length (mm)
Spherical Equivalent Refraction | 6 months, 12 months
  Evaluate change in Spherical Equivalent Refraction (Diopters) through manifest subjective refraction

CONTACTS AND LOCATIONS:
Locations (1):
- Essilor R&D Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bao J, Yang A, Huang Y, Li X, Pan Y, Ding C, Lim EW, Zheng J, Spiegel DP, Drobe B, Lu F, Chen H. One-year myopia control efficacy of spectacle lenses with aspherical lenslets. Br J Ophthalmol. 2022 Aug;106(8):1171-1176. doi: 10.1136/bjophthalmol-2020-318367. Epub 2021 Apr 2. PMID 33811039